CLINICAL TRIAL: NCT01215058
Title: Gastroprotective Agent Compliance in Patients at Risk Suffering From a Gastrointestinal Bleeding Ulcer or a Symptomatic Ulcer With Non-steroidal Anti-inflammatory Drug (NSAID) in France
Brief Title: Gastroprotective Agent Compliance in Patients at Risk Suffering From a Gastrointestinal(GI) Ulcer
Status: Withdrawn | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Marketing Company Medical Director, AstraZeneca
Other Study IDs: NIS-PFR-DUM-2010/2
Record Dates: First submitted 2010-09-28; First posted 2010-10-05 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Gastrointestinal Hemorrhage; Ulcer
Keywords: Compliance, France; Gastrointestinal bleeding ulcer or symptomatic ulcer with NSAID
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Ulcer; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to assess gastroprotective agent compliance in patients at risk suffering from a gastrointestinal bleeding ulcer or a symptomatic ulcer with NSAID.

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk suffering from a gastrointestinal bleeding ulcer or a symptomatic ulcer confirmed by endoscopy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital sample
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Gastroprotective agent compliance | At the end of 1 month

SECONDARY OUTCOMES:
Clinical characteristics of those ulcers with NSAID | At the end of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Bretagne, Study Chair — Service gastro-enterologie et hepatologieCHRU Pontchaillou35033 RENNES cedex France; Gerard Thiefin, Study Chair — Service Hepato-Gastroenterologie CHU Reims51092 REIMS cedex France; Genevieve BONNELYE, Principal Investigator — KantarHealth - France138, avenue Marx Dormoy92120 Montrouge cedex